CLINICAL TRIAL: NCT05624658
Title: Effect of Combined Lipid-lowering Therapy on Atherosclerotic Plaque Vulnerability in Patients With Acute Coronary Syndrome, a Prospective, Open-label, Randomized, Single-center Study
Brief Title: Effect of Combined Lipid-lowering Therapy on Atherosclerotic Plaque Vulnerability in Patients With ACS
Acronym: Combi-LLT ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samara Regional Cardiology Dispensary (Other)
Collaborators: Samara State Medical University (Other)
Responsible Party: Principal Investigator, Prof. Dmitry Duplyakov FESC, Medical Director, Samara Regional Cardiology Dispensary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SamaraRCD-1
Record Dates: First submitted 2022-11-08; First posted 2022-11-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dyslipidemias
Keywords: acute coronary syndrome; PCI; plaque vulnerability; combined lipid-lowering therapy; PCSK9 inhibitors; Ezetimibe; coronary artery computed tomography
MeSH Terms: conditions — Dyslipidemias; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Patients who did not reach the target LDL-C values 1 month after the development of ACS on the 2nd visit will be randomized into two groups of 60 patients each. Group 1 - taking PCSK9 inhibitors while taking Atorvastatin at a dose of 80 mg / day. Group 2 - receiving Ezetimibe at a dose of 10 mg in combination with Atorvastatin 80 mg / day. Also, on the 2nd visit, patients will undergo CCTA, an assessment of the CAVI index and a laboratory tests (blood count, lipid profile, ALAT, ASAT, Troponin I, Galectin -3, MMP -9, TIMP -1, high-sensitivity CRP, NGAL ). Every 3 months a visit is planned according to the schedule to monitor the effectiveness (blood count, ALAT, ASAT, lipid profile). Follow-up period will be 52 weeks, according to the schedule of visits. At the final visit, patients will undergo CCTA, assess the CAVI index and laboratory tests (blood count, lipid profile, Troponin I, Galectin-3, MMP-9, TIMP-1, high-sensitivity CRP, NGAL).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9 inhibitors in combination Atorvastatin at a dose of 80 mg /Rosuvastatin 40 mg/ day (Active Comparator): Patients who showed high compliance and did not reach the target LDL-C values 1 month after the development of ACS on the 2nd visit will be randomized into two groups of 60 patients each. Group 1 - taking PCSK9 inhibitors (Alirocumab 150 mg by subcutaneous injection once every 2 weeks or Evolocumab 140 mg by subcutaneous injection once every 2 weeks - open-label prescription of drugs) while taking Atorvastatin at a dose of 80 mg./ Rosuvastatin 40 mg / day.
  Interventions: Combination Product: Combined Lipid-lowering Therapy
- Ezetimibe at a dose of 10 mg in combination with Atorvastatin 80 mg / Rosuvastatin 40 mg/ day. (Active Comparator): Group 2 - receiving Ezetimibe at a dose of 10 mg in combination with Atorvastatin 80 mg / Rosuvastatin 40 mg/day.
  Interventions: Combination Product: Combined Lipid-lowering Therapy

INTERVENTIONS:
Combination Product: Combined Lipid-lowering Therapy — the effect of high-dose combined lipid-lowering therapy (statins+ezetimibe vs statins+PCSK9 inhibitors) on the vulnerability characteristics of atherosclerotic plaques assessed using multimodal imaging (coronary artery computed tomography and optical coherence tomography), as well as biomarkers in patients with acute coronary syndrome for 52 weeks.
  Other Names: invasive coronary angiography, coronary artery commputed tomography, OCT, CAVI index

SUMMARY:
The study is prospective, open-label, randomized, single-center study involving patients admitted on an emergency basis with an acute coronary syndrome (ACS) clinic who underwent PCI of an infarct-related artery (IRA) and had intermediate coronary artery lesions (50-70% stenosis diameter) and elevated LDL-C ( > 1.4 mmol/l) despite statin therapy at the highest dosage. Patients who showed high compliance and did not reach the target LDL-C values 1 month after the development of ACS on the 2nd visit will be randomized into two groups of 60 patients each. Group 1 - taking PCSK9 inhibitors (Alirocumab 150 mg by subcutaneous injection once every 2 weeks or Evolocumab 140 mg by subcutaneous injection once every 2 weeks - open-label prescription of drugs) while taking Atorvastatin at a dose of 80 mg / day. Group 2 - receiving Ezetimibe at a dose of 10 mg in combination with Atorvastatin 80 mg / day.

DETAILED DESCRIPTION:
The study will enroll 120 patients with ACS admitted on an emergency basis to the Hospital. All patients will undergo PCI of the infarct-related artery (IRA), as well as intracoronary imaging with OCT of one or two non-IRA. During hospitalization, patients will receive standard therapy of ACS according to clinical recommendations, while Atorvastatin will initially be prescribed at a maximum dosage of 80 mg / day. Patients who showed high compliance and did not reach the target LDL-C values 1 month after the development of ACS on the 2nd visit will be randomized into two groups of 60 patients each. Group 1 - taking PCSK9 inhibitors (Alirocumab 150 mg by subcutaneous injection once every 2 weeks or Evolocumab 140 mg by subcutaneous injection once every 2 weeks - open-label prescription of drugs) while taking Atorvastatin at a dose of 80 mg / day. Group 2 - receiving Ezetimibe at a dose of 10 mg in combination with Atorvastatin 80 mg / day.

Also, on the 2nd visit, patients will undergo coronary artery computed tomography (CCTA): assessment of the CAVI index and a laboratory tests (blood count, lipid profile, ALAT, ASAT, Troponin I, Galectin -3, MMP -9, TIMP -1, high-sensitivity CRP, NGAL ). Every 3 months a visit is planned according to the schedule to monitor the effectiveness (blood count, ALAT, ASAT, lipid profile).

Follow up duration will be 52 weeks, according to the schedule of visits. At the final visit, patients will undergo CCTA, CAVI index and laboratory tests (blood count, lipid profile, ALAT, ASAT, Troponin I, Galectin -3, MMP -9, TIMP -1, high-sensitivity CRP, NGAL).

ELIGIBILITY:
Inclusion Criteria:

* gender (any);
* age 18-75 years;
* admission < 24 hours after pain onset
* acute coronary syndrome with at least one coronary artery stenosis requiring PCI;
* one or two non-IRA (coronary artery lumen diameter according to CAG >20% and <50% and no need for revascularization within the next 6 months according to the investigator)
* not taking statins for at least 3 (6) months or not achieving the target level of LDL-C at admission
* failure to achieve the target level of LDL-C ≥1.4 mmol/l on the second visit;
* signed informed consent

Exclusion Criteria:

* previous MI
* history of revascularization (PCI/CABG)
* presence of non-IRA stenoses ≥50%.
* multivessel lesion, including significant stenosis of the LM
* EF < 40%,
* Killip III-IV.
* NYHA III-IV
* significant calcification or tortuosity of the coronary arteries, limiting OCT
* intolerance to statins, aspirin, P2Y12 inhibitors
* patients who have previously received PCSK9 inhibitors and/or Ezetimib
* treatment with systemic steroids or systemic cyclosporine within the last 3 months
* collagenoses and inflammatory diseases,
* oncological diseases within the last 5 years,
* scheduled surgery within 3 months
* persons suffering from mental disorders
* pregnancy, breastfeeding period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Percent of change plaque vulnerability parameters on CCTA data | 52 weeks
  change plaque vulnerability parameterson coronary artery computed tomography in non-IRA coronary arteries (positive remodeling; the presence of a low-density area in the plaque (less than 30 HU *); point calcifications in the composition of the plaque; ring-shaped enhancement of X-ray density along the periphery of the plaque, not exceeding 130 HU, or the phenomenon of "circular glow")

SECONDARY OUTCOMES:
The number of participants with death, stent thrombosis/restenosis, nonfatal MI, hospitalization due to unstable angina, revascularization within 1 year | 52 weeks
  assessment via telemedicine consultation every month and at follow-up visits every 3 months
Total cholesterol, LDL-C, HDL-C, triglycerides levels after 52 weeks | 52 weeks
  blood sampling at control visits every 3 months
dynamics of level hs-Troponin I within 1 year (ng/l) | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level hs-CRP within 1 year (mg/l) | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level NLR within 1 year | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level Galectin- 3 within 1 year (ng/ml) | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level MMP-9 within 1 year (ng/ml) | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level TIMP - 1 within 1 year (ng/ml) | 52 weeks
  blood sampling at the second visit and 12 months later
dynamics of level NGAL within 1 year (ng/ml) | 52 weeks
  blood sampling at the second visit and 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Duplyakov, Principal Investigator — Samara State Medical Universiry
Locations (1):
- Samara Regional Cardiology Dispansery, Samara, Russia

IPD SHARING:
Plan to Share IPD: No